CLINICAL TRIAL: NCT05613621
Title: Dissection of the Molecular and Immunological Interaction in Patients With Hepatocellular Carcinoma of Viral and Non-viral Etiologies
Brief Title: Dissection of the Molecular and Immunological Interaction in Patients With HCC of Viral and Non-viral Etiologies
Acronym: T4222
Status: Active, not recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Mackay Memorial Hospital (Other); National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: T4222
Record Dates: First submitted 2022-11-01; First posted 2022-11-14 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; next-generation sequencing; precision medicine
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — next-generation sequencing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training cohort: Consisting of 4 sub-groups: HBV (+) steatosis (+), HBV (-) steatosis (+), HBV (+) steatosis (-) and HBV (-) steatosis (-). HBV (+) is defined as either: (a) HBsAg (+) or (b) HBsAg (-) anti-HBc (+) and HBV DNA detectable in blood or tumor tissue. Steatosis is defined by histology. We will enroll 400 patients who had sufficient tissue for testing in the training cohort.
- validation cohort: For the validation cohort, the clinical and pathological information will be obtained retrospectively by TCOG and will take 6 months to identify eligible patients for the 4 sub-groups listed above.

SUMMARY:
This project will clarify the potential interaction between HBV infection and steatosis, and their impact on genetic alterations and tumor immune microenvironment.

DETAILED DESCRIPTION:
This study will start with a "training cohort" of the NTUH and NTU Cancer Center patients, consisting of 4 sub-groups: HBV (+) steatosis (+), HBV (-) steatosis (+), HBV (+) steatosis (-) and HBV (-) steatosis (-). HBV (+) is defined as either: (a) HBsAg (+) or (b) HBsAg (-) anti-HBc (+) and HBV DNA detectable in blood or tumor tissue. Steatosis is defined by histology. We will enroll 400 patients who had sufficient tissue for testing in the training cohort. The following studies will be performed: (1) NGS of targeted genes panel using the National Health Research Institutes precision medicine platform; (2) transcriptomic analysis of immune microenvironment using RNA-seq and multiplex immunofluorescence staining; (3) lipotoxic genotyping for SNPs; (4) clinical outcomes of MAFLD vs. non-MAFLD. The genetic and immunological features will be further tested by a "validation cohort", from collaborative hospitals. This project will clarify the potential interaction between HBV infection and steatosis, and their impact on genetic alterations and tumor immune microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female or male patients aged ≥20 years.
2. HCC has been histologically confirmed with resection specimen.
3. The surgery should be performed with curative intent after 2015 in the study hospital.
4. Availability of serum HBsAg and Anti-HBc data in the electronic medical record.
5. Availability of imaging data performed within 3 months before the surgery in the electronic medical record. (at least one of the following: computed tomography, magnetic resonance imaging, abdominal sonography).
6. Informed consent is obtained. Willingness to provide the residual operative slides and medical records.

Exclusion Criteria:

1. Fibrolamellar HCC, sarcomatoid HCC, or a mixture of cholangiocarcinoma and HCC
2. Exclusion of HCV patients (Anti-HCV positive)
3. Inability to cooperate by providing a complete medical history.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hepatocellular carcinoma patients
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
transcriptomic analysis of immune microenvironment | 2 Years
  using RNA-seq and multiplex immunofluorescence staining
lipotoxic genotyping for SNPs | 2 years
  lipotoxic genotyping for SNPs
clinical outcomes of MAFLD vs. non-MAFLD. | 2 years
  clinical outcomes of MAFLD vs. non-MAFLD.

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Wu Liu, Study Director — Taiwan Cooperative Oncology Group, NHRI
Locations (4):
- Taiwan (4):
  - National Cheng-Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - National Taiwan University Cancer Center, Taipei